CLINICAL TRIAL: NCT03824379
Title: The Impact of Magnesium Supplementation on the Clinical Outcome of Patients of Diabetic Nephropathy
Brief Title: Magnesium Supplementation in Diabetic Nephropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Nihal Mohamed Halawa, clinical Pharmacist, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHCL932
Record Dates: First submitted 2019-01-26; First posted 2019-01-31 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Diabetic Nephropathies
Keywords: magnesium; diabetic nephropathy; osteocalcin
MeSH Terms: conditions — Diabetic Nephropathies | interventions — magnesium citrate; Hypoglycemic Agents

STUDY DESIGN:
Intervention Model Description: prospective randomized controlled open label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Magnesium arm (Experimental): 30 patients will receive the standard therapy (anti-diabetic ) + magnesium supplement
  Interventions: Dietary Supplement: Magnesium citrate; Drug: Antidiabetic
- Control (Active Comparator): 30 patients will receive the standard therapy (anti-diabetic)
  Interventions: Drug: Antidiabetic

INTERVENTIONS:
Dietary Supplement: Magnesium citrate — magnesium citrate equivalent 20-30 mmol elemental magnesium
  Arms: Magnesium arm
Drug: Antidiabetic — insulin or oral hypoglycemics

SUMMARY:
Higher prevalence of hypomagnesaemia in diabetic patients with nephropathy was compared to those without nephropathy. Serum magnesium levels were significantly inversely correlated with serum creatinine and U-A/C ratio, and positively correlated with glomerular filtration rate (GFR).

Hence, Magnesium supplementation using magnesium salts could be a good approach to improve the cardiovascular complications, insulin resistance index, lipid profile and kidney function in diabetic nephropathy patients.

DETAILED DESCRIPTION:
Diabetic nephropathy is a serious kidney-related complication of type 1 diabetes and type 2 diabetes. It is also called diabetic kidney disease. Up to 40 percent of people with diabetes eventually develop kidney disease. Over time, elevated blood sugar associated with uncontrolled diabetes causes high blood pressure which in turn damages the kidneys by increasing kidney filtration pressure. Complications of diabetic nephropathy include heart and blood vessel disease (cardiovascular disease), fluid retention and hyperkalemia. Magnesium (Mg) is the fourth most abundant cation in the body and the second most important intracellular cation. It plays an essential role in biological systems as co-factor for more than 300 essential enzymatic reactions such as signal transduction, energy metabolism, vascular processes and bone metabolism. Normal serum Mg concentrations ranges from 0.7 to 1.1 mmol/L (1.4-2.0 mEq/L or 1.7-2.4 mg/dL). Outcome studies in the general population have indicated potential associations between low serum Mg levels and atherosclerosis, hypertension, diabetes, and left ventricular hypertrophy, as well as both CVD mortality and all-cause mortality. Low SMg levels (1.4-1.9 mg/dL; 0.58-0.78 mM) were independently associated with all-cause death in patients with prevalent CKD. Higher prevalence of hypomagnesaemia in diabetic patients with nephropathy compared to those without nephropathy. Serum magnesium levels were significantly inversely correlated with serum creatinine and U-A/C ratio, and positively correlated with glomerular filtration rate (GFR). Magnesium deficiency promotes hydroxyapatite formation and calcification of vascular smooth muscle cells . It is closely related to insulin resistance and metabolic syndrome. A lower Mg level is directly associated with a faster deterioration of renal function in T2DM patients. Moreover, hypomagnesemia is associated with the long-term micro- and macrovascular complications of T2DM. A dysregulation of mineral metabolism, reflected by altered levels of magnesium and FGF-23, correlates with an increased urinary albumin to creatinine ratio (UACR) in type 2 diabetic patients with CKD stages 2-4. Also, a link between hypomagnesemia and atherogenic dyslipidemia alterations exists; a significantly raised total cholesterol and LDL and non-HDL in patients with CKD are observed, suggesting a link to increased cardiovascular risk in CKD patients. Increasing magnesium levels could attenuate the cardiovascular risk derived from hyperphosphatemia, hence the CKD progression. Current literature suggests that Mg may have a protective effect on the CV system. Mg supplementation improves the insulin resistance index and beta-cell function, and decreases hemoglobin A1c levels in type 2 DM patients. In animal models of vascular calcification VC, dietary supplementation with magnesium results in marked reduction in VC and mortality, improved mineral metabolism, including lowering of PTH, as well as improvement in renal function. Hence, Magnesium supplementation using magnesium salts could be a good approach to improve the cardiovascular complications, insulin resistance index, lipid profile and kidney function in diabetic nephropathy patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Type I or II diabetic patientCKD stage 3 ( eGFR = 30 - 59 ml/min) or stage 4 ( eGFR 15-29 ml/min)
3. Proteinuria 30-300 mg/dl (microalbuminuria)
4. Low SMg levels (1.4-1.9 mg/dL; 0.58-0.78 mM) to normal (1.7-2.4 mg/dL; 0.7 -1.1 mmol/L; 1.4-2.0 mEq/L).
5. Life expectancy >12 months.
6. Women of child-bearing age should be using contraceptives as Hormonal contraceptive or Intra-uterine device.

Exclusion Criteria:

1. Kidney donor recipient.
2. Current treatment with Mg supplements.
3. Any condition impairing intestinal absorption of Mg (e.g: chronic pancreatitis, short bowel syndrome)
4. Active malignancy.
5. Pregnancy or breastfeeding.
6. Cardiac Arrythmias.
7. Allergy towards the Mg supplement.
8. Participation in other interventional trials.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Change of Human Serum Osteocalcin level | Change from baseline Human Serum Osteocalcin level at 12 weeks
  Evaluation of the extent of cardiovadcular events

SECONDARY OUTCOMES:
Serum Insulin | Samples will be measured at baseline and after 12 weeks
  Evaluation of Glycemic Status
The homeostasis model assessment-estimated insulin resistance (HOMA-IR) | Assessed at baseline and after 12 weeks
  (HOMA-IR), developed by Matthews et al. will be used to assess insulin resistance. The following formula will be used in its calculation: HOMA IR = (fasting glucose mg/dl × fasting insulin μU/ml)/22.5 × 18. A normal value was considered to be <2.5
Hemoglobin A1c level | Samples will be measured at baseline and after 12 weeks
  Evaluation of Glycemic Status
Fasting and Post Prandial Blood Sugar level | Samples will be measured at baseline and after 12 weeks
  Evaluation of Glycemic Status
Serum creatinine | Samples will be measured at baseline and after 12 weeks
  Evaluation of kidney function
Blood Urea Nitrogen Concentration | Samples will be measured at baseline and after 12 weeks
  Evaluation of kidney function
eGFR using the MDRD equation | Samples will be measured at baseline and after 12 weeks
  Evaluation of kidney function. GFR (mL/min/1.73 m2) = 175 × (Scr)-1.154 × (Age)-0.203 × (0.742 if female) × (1.212 if African American)
Serum Magnesium | Samples will be measured at baseline, 6 weeks and 12 weeks
  Evaluation of SMg level
Evaluation of Lipid profile | Samples will be measured at baseline and after 12 weeks
  Serum Low-density Lipoprotein Cholesterol (LDL-C), High-density Lipoprotein Cholesterol (HDL-C), Total Cholesterol, Triglycerides
Fatigue Assessment | Assessed at baseline and after 12 weeks
  Fatigue Assessment using Fatigue Severity Scale (FSS). It is a 9-item scale which measures the severity of fatigue and its effect on a person's activities and lifestyle in a variety of disorders.
  > 4 points indicates no fatigue 4 points or more indicates increasing fatigue
Quality of Life (QoL) Assessment: D-39 Questionnaire | Assessed at baseline and after 12 weeks
  Quality of Life (QoL) assessment using D-39 Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Nihal Halawa, Principal Investigator — Faculty of Pharmacy - Ain Shams University
Locations (1):
- Ain Shams University Hospitals, Cairo, Abbasseia, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Halawa N, Elsaid TW, El Wakeel LM, Shawki MA. Impact of magnesium supplementation on clinical outcome and disease progression of patients with diabetic nephropathy: a prospective randomized trial. Ther Adv Chronic Dis. 2023 Dec 12;14:20406223231214641. doi: 10.1177/20406223231214641. eCollection 2023. PMID 38107482